CLINICAL TRIAL: NCT05323396
Title: Impact of Parasitic Infections on Intestinal Epithelial Barrier and Immune Activation Among Persons Living With HIV in Lilongwe, Malawi
Brief Title: HIV And Parasitic Infection (HAPI) Study
Acronym: HAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-2553; D43TW009340 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: HIV Coinfection
Keywords: parasitic infection; chronic immune activation; HIV coinfection; Malawi; sCD14; sCD163; I-FABP; intestinal damage
MeSH Terms: conditions — HIV Infections; Parasitic Diseases | interventions — Albendazole; Praziquantel; Metronidazole

STUDY DESIGN:
Intervention Model Description: This trial is closest to a parallel trial, but different from most clinical trials in that the participants will not be randomized by the study team. The two groups will be determined based on the results of the initial sample collection. Those with a result positive for intestinal parasitic infection (by either stool microscopy or stool PCR) will be in the "parasite-positive" group for the remainder of the study. Those negative for all of these will be in the "parasite-negative" group. The markers sCD14, sCD163, and I-FABP will be compared between the two groups. Additionally a comparison will be made between the pre-treatment and post-treatment levels of the "parasite-positive" participants.
Masking Description: The participants and the study team will know the results of the tests, and thus will know the groups that the participants are in, since only the "parasite-positive" participants will receive treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parasite-positive arm (Active Comparator): Participants will be evaluated for intestinal parasitic infection by stool microscopy or stool PCR. If positive by either of these, the participant will be treated for the detected parasitic infection. The biomarker levels of this parasite-positive group will be compared to the parasite-negative group. Additionally the parasite-positive pre-treatment biomarker levels will be compared to the parasite-positive post-treatment levels.
  Interventions: Drug: Antiparasitic medication
- Parasite-negative arm (No Intervention): Participants will be evaluated for intestinal parasitic infection by stool microscopy or stool PCR. If negative by all of these tests on the initial sample collection, the participants will not receive treatment and will be in the "parasite-negative"/no intervention arm.

INTERVENTIONS:
Drug: Antiparasitic medication — Participants in the "parasite-positive" group (based on positive result of either stool microscopy or stool PCR) will be administered antiparasitic treatment. Antiparasitic medication administered will be targeted to treat the parasite identified. See detailed description of protocol for medication, dose, and frequency that will be given for each parasitic infection identified.
  Participants with negative stool microscopy and negative stool PCR will not be administered treatment, thus will serve as controls.
  Other Names: Albendazole; Praziquantel; Metronidazole
  Arms: Parasite-positive arm

SUMMARY:
The overall goal of this study is to determine if periodic de-worming of persons living with HIV in intestinal parasite-endemic regions will lead to decreased morbidity and mortality associated with HIV by reducing immune activation and intestinal damage associated with these diseases. The hypothesis for this project is that intestinal parasitic infections contribute to a modifiable pro-inflammatory state in persons living with HIV (PLWH).

Aim 1: Determine the prevalence of intestinal parasitic infections in PLWH receiving care at an HIV-treatment center in Lilongwe, Malawi using a highly sensitive multi-parallel stool PCR test. Hypothesis: highly sensitive stool PCR testing will demonstrate that disease burden of parasitic infection in PLWH in Malawi is higher than historically reported based on stool microscopy.

Aim 2: Determine the impact of parasitic infection on intestinal damage and immune activation by measuring sCD14, sCD163, and intestinal fatty acid binding protein (I-FABP) in PLWH. Hypothesis: plasma biomarkers reflecting intestinal damage and immune activation are elevated in those with HIV and parasitic co-infection compared with parasite-negative participants with HIV.

Aim 3: Determine the impact of eradication of parasitic infection on intestinal damage and immune activation by measuring sCD14, sCD163, and intestinal fatty acid binding protein (I-FABP) in PLWH before and after treatment of parasitic co-infection. Hypothesis: plasma biomarkers reflecting intestinal damage and immune activation are elevated in those with HIV and parasitic co-infection, and these biomarkers decrease with anti-parasitic treatment.

DETAILED DESCRIPTION:
This is a prospective study in which participants will be enrolled in outpatient HIV clinics associated with Kamuzu Central Hospital in Lilongwe, Malawi, where there are over 25,000 patients in care with over 90% virally suppressed on ART.

Any subject meeting inclusion criteria and lacking exclusion criteria who is currently receiving care at the clinics affiliated with Kamuzu Central Hospital or Bwaila Hospital will be eligible to participate in this study. After informed consent is signed, a total of 10ml of blood, 20g stool sample, and 20mL urine sample will be collected. Each participant will be asked a series of questions. Clinical variables including age, sex, CD4+ T-cell count, and CD4% will be collected from the participant's medical chart.

Stool samples will be processed by stool microscopy in the local UNC Project Malawi laboratory, and the remaining sample will be stored at -80 degrees Celsius (C) until transported to the Laboratory of Parasitology National School of Tropical Medicine Baylor College of Medicine in Houston, Texas for detection of 9 different parasites and quantification of parasite burden by stool qPCR. Blood samples will be collected in EDTA-blood collection tubes and centrifuged. Plasma will be frozen at -80 degrees C at UNC Project Malawi until transport to the National School of Tropical Medicine Baylor College of Medicine for determination of levels of immune activation and gut mucosal impairment (sCD14, sCD163, and I-FABP). Urine samples will be evaluated by microscopy to look for Schistosoma haematobium at UNC Project Malawi laboratory.

Multi-parallel real-time quantitative PCR (qPCR) performed on stool will evaluate for 9 different parasites including Ascaris lumbricoides, Ancylostoma duodenale, Necator americanus, Schistosoma mansonii, Strongyloides stercoralis, Taenia solium, Trichuris trichiura, Entamoeba histolytica, and Giardia lamblia.

Participants that test positive for parasitic infection will be contacted and appropriate treatment administered according to the local standard of care. Albendazole single 400mg dose will be given for infection with Ascaris lumbricoides, Ancylostoma duodenale, Necator americanus, Trichuris trichiura. Albendazole 400mg daily for 5 days will be given for Strongyloides stercoralis. Praziquantel single dose 40mg/kg will be given for infection with Schistosoma mansoni and Schistosoma haematobium. Praziquantel single dose 10mg/kg will be given to treat intestinal infection with Taenia solium. Metronidazole 500mg two times a day x5 days for Giardia lamblia and 500mg three times a day x7 days for Entamoeba histolytica.

Follow up appointments will be performed 8-12 weeks after treatment and will include repeated blood and stool sample collection.

The study team anticipates enrollment of 120 patients in a period of 8-12 weeks. With an estimated intestinal parasite prevalence of 30%, the study team predicts 30 cases and 70 controls will be enrolled. Participants found to be positive at both the initial and follow up visit will be considered reinfected rather than treatment failure. These will be included in the analysis of prevalence, but the change in markers of immune activation will not be measured in this group since parasite clearance not established. Using Student's unpaired t-test to compare mean values of biomarkers between study groups, there will be 80% power to detect a difference of 0.434 x106 pg/ml, 0.56 mg/l, and 598 pg/ml between groups for biomarkers sCD14, sCD163, and I-FABP, respectively with effect sizes within the range of prior studies. Using paired t-tests to compare pre- and post-treatment biomarker levels, there will be 80% power to detect post-treatment changes of 0.317 x106/ml, 0.41 mg/l, and 435 pg/ml in sCD14, CD163, and I-FABP respectively.

Clinical variables including age, sex, and most recent CD4 count will be recorded. Clinical predictors of parasitic infection (eg CD4%) will be determined using multivariable logistical regression. Univariable linear regression will be used to determine associations between markers of immune activation (continuous outcome variable) and predictors including the clinical variables above as well as presence of multiple parasitic infections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* currently living in Malawi
* HIV-1 infection
* on ART ≥ 1 year with undetectable HIV RNA level at the last evaluation
* willingness to be treated with anti-parasitic therapy if infection with intestinal parasite is identified.

Exclusion Criteria:

* Use of antibiotics other than prophylaxis with trimethoprim-sulfamethoxazole within 60 days of screening
* Use of antiparasitic medication (ex- albendazole, praziquantel, metronidazole) in the last year
* Inflammatory bowel disease
* Gastrointestinal tract malignancy
* Major intestinal surgery during prior 2 years
* Coinfection with Mycobacterium tuberculosis
* Pregnancy, breastfeeding mother, or planning pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Reimer-McAtee, MD, Principal Investigator — University of North Carolina
Locations (1):
- Lighthouse Clinic, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: beginning 9 and continuing 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Sandler NG, Wand H, Roque A, Law M, Nason MC, Nixon DE, Pedersen C, Ruxrungtham K, Lewin SR, Emery S, Neaton JD, Brenchley JM, Deeks SG, Sereti I, Douek DC; INSIGHT SMART Study Group. Plasma levels of soluble CD14 independently predict mortality in HIV infection. J Infect Dis. 2011 Mar 15;203(6):780-90. doi: 10.1093/infdis/jiq118. Epub 2011 Jan 20. PMID 21252259
- [Background] Knudsen TB, Ertner G, Petersen J, Moller HJ, Moestrup SK, Eugen-Olsen J, Kronborg G, Benfield T. Plasma Soluble CD163 Level Independently Predicts All-Cause Mortality in HIV-1-Infected Individuals. J Infect Dis. 2016 Oct 15;214(8):1198-204. doi: 10.1093/infdis/jiw263. Epub 2016 Jun 28. PMID 27354366
- [Background] Cheru LT, Park EA, Saylor CF, Burdo TH, Fitch KV, Looby S, Weiner J, Robinson JA, Hubbard J, Torriani M, Lo J. I-FABP Is Higher in People With Chronic HIV Than Elite Controllers, Related to Sugar and Fatty Acid Intake and Inversely Related to Body Fat in People With HIV. Open Forum Infect Dis. 2018 Nov 5;5(11):ofy288. doi: 10.1093/ofid/ofy288. eCollection 2018 Nov. PMID 30515430

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After signing informed consent, participants provide laboratory samples for evaluation of parasitic infection.
Groups:
- Parasite-positive Arm: Participants will be evaluated for intestinal parasitic infection by stool microscopy, stool polymerase chain reaction (PCR) and Strongyloides IgG from plasma. If positive by either of these, the participant will be treated for the detected parasitic infection. The biomarker levels of this parasite-positive group will be compared to the parasite-negative group. Additionally the parasite-positive pre-treatment biomarker levels will be compared to the parasite-positive post-treatment levels.
  Antiparasitic medication: Participants in the "parasite-positive" group (based on positive result of either stool microscopy, stool PCR, or Strongyloides IgG) will be administered antiparasitic treatment. Antiparasitic medication administered will be targeted to treat the parasite identified. See detailed description of protocol for medication, dose, and frequency that will be given for each parasitic infection identified.
  Participants with stool microscopy, stool PCR, and Strongyloides IgG all negative will not be administered treatment, thus will serve as controls.
- Parasite-negative Arm: Participants will be evaluated for intestinal parasitic infection by stool microscopy, stool PCR and Strongyloides IgG from plasma. If negative by all of these tests on the initial sample collection, the participants will not receive treatment and will be in the "parasite-negative"/no intervention arm.
Period: Overall Study
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
Started | 36 | 84
Laboratory Evaluation Performed | 36 | 84
Received Intervention | 35 | 0
Completed | 34 | 49
Not Completed | 2 | 35
Not completed — Lost to Follow-up | 1 | 35
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Parasite-positive Arm: Participants will be evaluated for intestinal parasitic infection by stool microscopy, stool PCR and Strongyloides IgG from plasma. If positive by either of these, the participant will be treated for the detected parasitic infection. The biomarker levels of this parasite-positive group will be compared to the parasite-negative group. Additionally the parasite-positive pre-treatment biomarker levels will be compared to the parasite-positive post-treatment levels.
  Antiparasitic medication: Participants in the "parasite-positive" group (based on positive result of either stool microscopy, stool PCR, or Strongyloides IgG) will be administered antiparasitic treatment. Antiparasitic medication administered will be targeted to treat the parasite identified. See detailed description of protocol for medication, dose, and frequency that will be given for each parasitic infection identified.
  Participants with stool microscopy, stool PCR, and Strongyloides IgG all negative will not be administered treatment, thus will serve as controls.
- Total: Total of all reporting groups
Arm/Group | Parasite-positive Arm | Parasite-negative Arm | Total
Number analyzed (Participants) | 36 | 84 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [35 to 50] | 44 [38 to 50] | 43.5 [38 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 44 | 62
  Male | 18 | 40 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 84 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 84 | 120
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 36 | 84 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without Intestinal Parasitic Infection
Description: The number of participants with and without parasitic infection was determined based on diagnostic tests utilized. Participants with a positive result by either stool microscopy or stool PCR were considered "parasite-positive". Participants negative by both diagnostic tests were considered "parasite-negative".
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Participants With and Without Parasitic Infection: Participants evaluated for intestinal parasitic infection by stool microscopy, stool PCR and Strongyloides IgG from plasma. If positive by either of these, the participant was treated for the detected parasitic infection.
Arm/Group | Participants With and Without Parasitic Infection
Number analyzed (Participants) | 120
Participants
  Parasite-positive | 36
  Parasite-negative | 84

2. Primary Outcome: Mean Soluble CD14 (sCD14) Levels
Description: The level of sCD14 detected in plasma will be measured in all patients at the baseline visit. The mean level of sCD14 of the parasite-positive group will be compared to the mean level of sCD14 of the parasite-negative group (µg/mL) using Student's unpaired t-test.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
Number analyzed (Participants) | 36 | 84
µg/mL | 1.42 (0.39) | 1.52 (0.42)
Statistical Analysis 1: Comparison: Parasite-positive Arm vs Parasite-negative Arm; Test type: Other; p = 0.19, Student's unpaired t-test

3. Primary Outcome: Mean Soluble CD163 (sCD163) Levels
Description: The level of sCD163 detected in plasma will be measured in all patients at the baseline visit. The mean level of sCD163 of the parasite-positive group will be compared to the mean level of sCD163 of the parasite-negative group (ng/mL) using Student's unpaired t-test.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
Number analyzed (Participants) | 36 | 84
ng/mL | 736.13 (212.63) | 744.61 (218.06)
Statistical Analysis 1: Comparison: Parasite-positive Arm vs Parasite-negative Arm; Test type: Other; p = 0.85, Student's unpaired t-test

4. Primary Outcome: Mean Intestinal Fatty-acid Binding Protein (I-FABP) Levels
Description: The level of I-FABP detected in plasma will be measured in all patients at the baseline visit. The mean level of I-FABP of the parasite-positive group will be compared to the mean level of I-FABP of the parasite-negative group (ng/mL) using Student's unpaired t-test.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
Number analyzed (Participants) | 36 | 84
ng/mL | 3.33 (3.22) | 3.49 (2.62)
Statistical Analysis 1: Comparison: Parasite-positive Arm vs Parasite-negative Arm; Test type: Other; p = 0.77, Student's unpaired t-test

5. Primary Outcome: Percent Change of sCD14 Levels Pre- and Post-treatment
Description: The level of sCD14 detected in plasma will be measured in all patients at the initial visit and the follow-up visit (µg/mL). The percent change of sCD14 from pre-treatment to post-treatment levels of the parasite-positive group will be compared to the percent change of sCD14 from pre- to post-treatment levels of the parasite-negative participants.
Time Frame: Baseline, 6 months after baseline visit
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
Number analyzed (Participants) | 34 | 49
percent change | 8.52 (30.41) | -0.90 (24.36)
Statistical Analysis 1: Comparison: Parasite-positive Arm vs Parasite-negative Arm; Test type: Other; p = 0.12, student's unpaired t-test

6. Primary Outcome: Percent Change of sCD163 Levels Pre- and Post-treatment
Description: The level of sCD163 detected in plasma will be measured in all patients at the initial visit and the follow-up visit (ng/mL). The percent change of sCD163 from pre-treatment to post-treatment levels of the parasite-positive group will be compared to the percent change of sCD163 from pre- to post-treatment levels of the parasite-negative participants.
Time Frame: Baseline, 6 months after baseline visit
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
Number analyzed (Participants) | 34 | 49
percent change | -7.38 (15.18) | -8.56 (24.71)
Statistical Analysis 1: Comparison: Parasite-positive Arm vs Parasite-negative Arm; Test type: Other; p = 0.81, student's unpaired t-test

7. Primary Outcome: Percent Change of I-FABP Levels Pre- and Post-treatment
Description: The level of I-FABP detected in plasma will be measured in all patients at the initial visit and the follow-up visit (ng/mL). The percent change of I-FABP levels from pre-treatment to post-treatment of the parasite-positive group will be compared to the percent change of I-FABP levels pre- and post-treatment of the parasite-negative participants.
Time Frame: Baseline, 6 months after baseline visit
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
Number analyzed (Participants) | 34 | 49
percent change | 79.85 (268.28) | 107.31 (278.19)
Statistical Analysis 1: Comparison: Parasite-positive Arm vs Parasite-negative Arm; Test type: Other; p = 0.65, student's unpaired t-test

ADVERSE EVENTS:
Time Frame: From receipt of intervention through the 3-month follow-up, a total of 3 months
Description: Since the parasite negative arm did not receive an intervention, adverse events were not collected for this arm.
Arm/Group | Parasite-positive Arm | Parasite-negative Arm
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/0
Other Adverse Events (participants affected / at risk) | 0/36 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT05323396/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT05323396/ICF_000.pdf